CLINICAL TRIAL: NCT06113016
Title: A Phase II Randomized Placebo-Controlled Study of Fisetin and Exercise to Prevent Frailty in Breast Cancer Survivors
Brief Title: Prevention of Frailty With Fisetin and Exercise in Breast Cancer Survivors
Acronym: PROFFi
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Jonsson Comprehensive Cancer Center (Other)
Collaborators: National Institutes of Health (NIH) (NIH); National Cancer Institute (NCI) (NIH); Rising Tide Foundation (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Supportive Care
Other Study IDs: 23-001171; P30CA016042 (NIH); R01CA280088 (NIH); NCI-2023-06774 (Registry Identifier: CTRP (Clinical Trial Reporting Program))
Record Dates: First submitted 2023-10-26; First posted 2023-11-02 (Actual); Last update posted 2025-07-08 (Actual); Status verified 2025-06

CONDITIONS: Anatomic Stage I Breast Cancer American Joint Committee on Cancer (AJCC) v8; Anatomic Stage II Breast Cancer AJCC v8; Anatomic Stage III Breast Cancer AJCC v8; Early Stage Breast Carcinoma
MeSH Terms: interventions — Specimen Handling; Early Intervention, Educational; Educational Status; Methods; fisetin; Exercise Test

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: This is a double-blind study with respect to study agent. Because participants cannot be blinded to exercise training, the outcomes assessor (but not the physicians or participants) will be blinded to the training status of participants.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (4):
- Arm A (fisetin, physical activity handout) (Active Comparator): Patients receive fisetin PO on days 1-3 of each cycle. Treatment repeats every 14 days for 8 cycles in the absence of disease progression or unacceptable toxicity. Patients also receive handout on the importance of physical activity during baseline. Patients undergo collection of blood samples on study.
  Interventions: Procedure: Biospecimen Collection; Other: Educational Intervention; Drug: Fisetin; Other: Physical Performance Testing; Other: Quality-of-Life Assessment; Other: Questionnaire Administration
- Arm AB (fisetin, tailored exercise training) (Experimental): Patients receive fisetin PO on days 1-3 of each cycle. Treatment repeats every 14 days for 8 cycles in the absence of disease progression or unacceptable toxicity. Patients also receive individually tailored supervised exercise training consisting of 30-45 minutes of aerobic training and 20-30 minutes of resistance training three times a week over 16 weeks. Patients undergo collection of blood samples on study.
  Interventions: Procedure: Biospecimen Collection; Other: Exercise Intervention; Drug: Fisetin; Other: Physical Performance Testing; Other: Quality-of-Life Assessment; Other: Questionnaire Administration
- Arm B (placebo, tailored exercise training) (Active Comparator): Patients receive placebo PO on days 1-3 of each cycle. Treatment repeats every 14 days for 8 cycles in the absence of disease progression or unacceptable toxicity. Patients also receive individually tailored supervised exercise training consisting of 30-45 minutes of aerobic training and 20-30 minutes of resistance training three times a week over 16 weeks. Patients undergo collection of blood samples on study.
  Interventions: Procedure: Biospecimen Collection; Other: Exercise Intervention; Other: Physical Performance Testing; Drug: Placebo Administration; Other: Quality-of-Life Assessment; Other: Questionnaire Administration
- Arm C (placebo, physical activity handout) (Active Comparator): Patients receive placebo PO on days 1-3 of each cycle. Treatment repeats every 14 days for 8 cycles in the absence of disease progression or unacceptable toxicity. Patients also receive handout on the importance of physical activity during baseline. Patients undergo collection of blood samples on study.
  Interventions: Procedure: Biospecimen Collection; Other: Educational Intervention; Other: Physical Performance Testing; Drug: Placebo Administration; Other: Quality-of-Life Assessment; Other: Questionnaire Administration

INTERVENTIONS:
Procedure: Biospecimen Collection — Undergo collection of blood samples
  Other Names: Biological Sample Collection; Biospecimen Collected; Specimen Collection
Other: Educational Intervention — Receive handout on physical activity
  Other Names: Education for Intervention; Intervention by Education; Intervention through Education; Intervention, Educational
  Arms: Arm A (fisetin, physical activity handout); Arm C (placebo, physical activity handout)
Other: Exercise Intervention — Receive individually tailored exercise intervention
  Arms: Arm AB (fisetin, tailored exercise training); Arm B (placebo, tailored exercise training)
Drug: Fisetin — Given PO
  Other Names: 3,3',4',7-Tetrahydroxyflavone; 7,3',4'-Flavon-3-ol
  Arms: Arm A (fisetin, physical activity handout); Arm AB (fisetin, tailored exercise training)
Other: Physical Performance Testing — Ancillary studies
  Other Names: Physical Fitness Testing; Physical Function Testing
Drug: Placebo Administration — Given PO
  Arms: Arm B (placebo, tailored exercise training); Arm C (placebo, physical activity handout)
Other: Quality-of-Life Assessment — Ancillary studies
  Other Names: Quality of Life Assessment
Other: Questionnaire Administration — Ancillary studies

SUMMARY:
This phase II trial tests how well fisetin and exercise works in preventing frailty in breast cancer survivors. Fisetin is a natural substance found in strawberries and other foods and is available as a nutritional supplement. Nutritional supplements may be useful in eliminating cells that have undergone a process called senescence. Senescence is when a cell ages and permanently stops dividing but does not die. Over time, large numbers of these cells build up in tissues throughout the body and can release harmful substances that cause inflammation and damage nearby healthy cells. Giving fisetin may eliminate senescent cells in patients with breast cancer undergoing physical activity.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVE:

I. To determine the effect of fisetin and/or exercise on physical function, as assessed using the 6-minute walk distance (6MWD), in chemotherapy-treated postmenopausal breast cancer survivors.

SECONDARY OBJECTIVES:

I. To determine the effect of fisetin and/or exercise on heart rate and step count, as measured by wearable device.

II. To determine the effect of fisetin on other measures of physical function beyond 6MWD (short physical performance battery [SPPB], grip strength, frailty phenotype, physical activity).

III. To determine the effect of fisetin and/or exercise on fatigue (Borg Rating of Perceived Exertion [RPE]).

IV. To determine the effect of fisetin and/or exercise on neuropathy (Quality of Life Questionnaire - Chemotherapy-Induced Peripheral Neuropathy 20 [QLQ-CIPN20]).

V. To determine the effect of fisetin and/or exercise on cognition (Patient Reported Outcomes Measurement Information System [PROMIS] cognitive function short form).

VI. To determine the effect of fisetin and/or exercise on health-related quality of life (Short Form [SF]-36).

VII. To determine the effect of fisetin on local and distant recurrence free survival (RFS).

VIII. To determine the effect of fisetin on breast cancer-specific survival and overall survival.

IX. To evaluate the safety and tolerability (National Cancer Institute [NCI] Common Terminology Criteria for Adverse Events [CTCAE] version [v]5.0) of fisetin.

X. To estimate rates of adherence to fisetin and/or exercise regimen.

EXPLORATORY OBJECTIVES:

I. To determine the effect of fisetin and/or exercise on p16 expression in peripheral CD3+ T-cells.

II. To determine the effect of fisetin and/or exercise on circulating senescence-associated secretory phenotype (SASP) inflammatory factors in blood and urine.

OUTLINE: Patients are randomized to 1 of 4 arms.

ARM AB: Patients receive fisetin orally (PO) on days 1-3 of each cycle. Treatment repeats every 14 days for 8 cycles in the absence of disease progression or unacceptable toxicity. Patients also receive individually tailored supervised exercise training consisting of 30-45 minutes of aerobic training and 20-30 minutes of resistance training three times a week over 16 weeks. Patients undergo collection of blood samples on study.

ARM A: Patients receive fisetin PO on days 1-3 of each cycle. Treatment repeats every 14 days for 8 cycles in the absence of disease progression or unacceptable toxicity. Patients also receive handout on the importance of physical activity during baseline. Patients undergo collection of blood samples on study.

ARM B: Patients receive placebo PO on days 1-3 of each cycle. Treatment repeats every 14 days for 8 cycles in the absence of disease progression or unacceptable toxicity. Patients also receive individually tailored supervised exercise training consisting of 30-45 minutes of aerobic training and 20-30 minutes of resistance training three times a week over 16 weeks. Patients undergo collection of blood samples on study.

ARM C: Patients receive placebo PO on days 1-3 of each cycle. Treatment repeats every 14 days for 8 cycles in the absence of disease progression or unacceptable toxicity. Patients also receive handout on the importance of physical activity during baseline. Patients undergo collection of blood samples on study.

Following completion of study intervention, patients are followed up on days 120 and 180 and then annually for up to 3 years.

ELIGIBILITY:
Inclusion Criteria:

* Women who are postmenopausal at the start of study treatment

  * Postmenopausal status will be established as follows: Women who are 50 years or older and who are not menstruating for greater than 12 months will be considered postmenopausal. Women who are less than 50 years with an intact uterus and ovaries must have chemically induced menopause (e.g., ovarian suppression) to be considered postmenopausal
* Women with a diagnosis of early-stage breast cancer (stage I, II, III) treated with neo/adjuvant chemotherapy within 12 months of starting study treatment
* No evidence of active/recurrent breast cancer or other serious chronic illnesses
* Have evidence of pre-frail health, defined as a 6-minute walk distance (400-480m) at baseline
* Platelets > 60,000/mm^3
* White blood cell count > 2,000/mm^3
* Absolute neutrophil count > 500/mm^3
* Hemoglobin ≥ 8.0 g/dL
* Total bilirubin ≤ 3.0 X upper limit of normal (ULN)
* Aspartate aminotransferase (AST) ≤ 4.0 x ULN
* Alanine aminotransferase (ALT) ≤ 4.0 x ULN
* Estimated glomerular filtration rate (eGFR) of ≥ 30mL/min/1.73m^2 per the Modification of Diet in Renal Disease (MDRD) calculation. GFR (mL/min/1.73 m²) = 175 × (Scr)-1.154 × (Age)-0.203 × (0.742 if female) × (1.212 if African American)
* Ability to understand and the willingness to sign a written informed consent document

Exclusion Criteria:

* Cancer-directed chemotherapy, biological therapy, or immunotherapy within 30 days prior to the start of study treatment. Exceptions include: trastuzumab, pertuzumab, pembrolizumab, tamoxifen, and aromatase inhibitors
* Surgery and/or radiation within the last 30 days of starting study treatment (Exception: invasive non-major procedures such as an outpatient biopsy)
* Subjects taking medications that are considered prohibited

  * Exception: Subjects taking any of the medications under "Temporary medication adjustment required" may participate if they are otherwise eligible AND the medication can be safely withheld (from immediately before the 1st study agent administration until at least 10 hours after the last study agent administration, for each dosing interval)
* On herbal and natural medications with possible senolytic properties (i.e., curcumin, kava kava, St. John's wort) and are unable or unwilling to hold its administration 2 days prior to and during study treatment dosing. Exceptions include cannabidiol (CBD), vitamins, probiotics, and fish oil. Other herbal and natural medications may be permitted or prohibited per clinician discretion
* Subjects taking potentially senolytic agents within the last year: fisetin, quercetin, luteolin, dasatinib or imatinib (or other tyrosine kinase inhibitors), piperlongumine, or navitoclax
* Subjects on therapeutic doses of anticoagulants (e.g., warfarin, heparin, low molecular weight heparin, factor Xa inhibitors, etc.)
* Issues with tolerating oral medication (such as but not limited to, inability to swallow pills (gastrostomy [g]-tubes not allowed), malabsorption issues, ongoing nausea or vomiting during screening, history of Crohn's, gastric bypass/reduction, or celiac disease)
* Any other condition that would, in the investigator's judgment, contraindicate the patient's participation in the clinical study due to safety concerns with clinical study procedures
* Currently participating in another intervention research study seeking to improve functional status, alleviate frailty, muscle strength, exhaustion/fatigue, or cognitive function

Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 164 (Estimated)
Dates: Start 2024-07-23 (Actual); Primary Completion 2028-06-30 (Estimated); Study Completion 2028-12-30 (Estimated)

PRIMARY OUTCOMES:
Change in 6 minute walk distance (6MWD) | From baseline to day 120
  The 6MWD will assess the distance walked over 6 minutes and is measured in meters. A linear model will be fit to outcome variable (change score) with a factor variable representing the four study arms and control for baseline 6MWD, site, and age stratum. The analysis will be conducted as intention-to-treat analysis. Will conduct an as-treated analysis, comparing the treatments received (instead of as-randomized).

SECONDARY OUTCOMES:
Change in heart rate | From baseline to day 120
  Changes will be calculated for treatments A, B, AB, and C. Linear models will be used to determine treatment effects using the two-stage testing procedure. Will conduct as-treated analysis and linear mixed models will also be fit to examine trends.
Change in step count | From baseline to day 120
  Changes will be calculated for treatments A, B, AB, and C. Linear models will be used to determine treatment effects using the two-stage testing procedure. Will conduct as-treated analysis and linear mixed models will also be fit to examine trends.
Change in short physical performance battery (SPPB) | From baseline to day 120
  Changes will be calculated for treatments A, B, AB, and C. Linear models will be used to determine treatment effects using the two-stage testing procedure. Will conduct as-treated analysis and linear mixed models will also be fit to examine trends.
Change in grip strength | From baseline to day 120
  Changes will be calculated for treatments A, B, AB, and C. Linear models will be used to determine treatment effects using the two-stage testing procedure. Will conduct as-treated analysis and linear mixed models will also be fit to examine trends.
Change in frailty phenotype | From baseline to day 120
  Changes will be calculated for treatments A, B, AB, and C. Linear models will be used to determine treatment effects using the two-stage testing procedure. Will conduct as-treated analysis and linear mixed models will also be fit to examine trends.
Change in physical function subsection of Short Form (SF)-36 | From baseline to day 120
  Changes will be calculated for treatments A, B, AB, and C. Linear models will be used to determine treatment effects using the two-stage testing procedure. Will conduct as-treated analysis and linear mixed models will also be fit to examine trends.
Change in the Borg Rating of Perceived Exertion (RPE) | From baseline to day 120
  Changes will be calculated for treatments A, B, AB, and C. Linear models will be used to determine treatment effects using the two-stage testing procedure. Will conduct as-treated analysis and linear mixed models will also be fit to examine trends.
Change in Quality of Life Questionnaire - Chemotherapy-Induced Peripheral Neuropathy 20 (QLQ-CIPN20) scores | From baseline to day 120
  Changes will be calculated for treatments A, B, AB, and C. Linear models will be used to determine treatment effects using the two-stage testing procedure. Will conduct as-treated analysis and linear mixed models will also be fit to examine trends. Quality of Life Questionnaire - Chemotherapy-Induced Peripheral Neuropathy 20 (QLQ-CIPN20). Scoring range is from 20-80. A lower score defines a more favorable outcome.
Change in Patient Reported Outcomes Measurement Information System (PROMIS) cognitive function short form score | From baseline to day 120
  Changes will be calculated for treatments A, B, AB, and C. Linear models will be used to determine treatment effects using the two-stage testing procedure. Will conduct as-treated analysis and linear mixed models will also be fit to examine trends. Patient Reported Outcomes Measurement Information System (PROMIS) cognitive function short form. A composite score of 0-40 is created with higher scores indicating a better health outcome.
Change in SF-36 scores | From baseline to day 120
  Changes will be calculated for treatments A, B, AB, and C. Linear models will be used to determine treatment effects using the two-stage testing procedure. Will conduct as-treated analysis and linear mixed models will also be fit to examine trends. Soring range is 0-100. a higher score defines a more favorable outcome.
Local and distant recurrence free survival | Up to 3 years
Breast cancer specific survival | Up to 3 years
Overall survival | Up to 3 years
Incidence of adverse events | Up to day 120
  Measured by National Cancer Institute (NCI) Common Terminology Criteria for Adverse Events (CTCAE) version (v)5.0.
Adherence rate | Up to day 120
  Treatment adherence will be evaluated in clinic on day 1 of each cycle and via telephone follow-up on day 2, day 3 of each cycle. Adherence information obtained will include the start and finish time for ingesting the drug and the number of pills ingested. Adherence will also be collected in a pill diary.

CONTACTS AND LOCATIONS:
Overall Officials: Mina S Sedrak, Principal Investigator — UCLA / Jonsson Comprehensive Cancer Center
Locations (6):
- United States (6):
  - UCLA Health Cancer Care in Alhambra, Alhambra, California
  - UCLA Health Beverly Hills Primary & Specialty Care, Beverly Hills, California
  - UCLA Health Burbank Primary & Specialty Care, Burbank, California
  - UCLA / Jonsson Comprehensive Cancer Center, Los Angeles, California
  - UCLA Health Primary Care in Marina del Rey, Marina del Rey, California
  - UCLA Health Primary Care in Pasadena, Pasadena, California